CLINICAL TRIAL: NCT03655119
Title: Psychiatric Emergency Services Family Support and Follow-Up Program
Brief Title: PES Family Support and Follow-Up Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was paused due to COVID-19 restrictions related to recruitment and will not resume.
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other); Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cynthia Ewell Foster, Clinical Assistant Professor, University of Michigan
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00125065; 5U79SM061767 (SAMHSA)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Suicide
Keywords: Child; Adoelscent; Crisis Intervention
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): Youth and parents will complete surveys at index PES visit regarding suicide related risk and protective factors. Parents and youth will complete a follow-up survey at 3 days (parents only) and 2 weeks (parents and youth) post discharge. At 3 days and 2 weeks, parents will complete a survey that evaluates adherence to safety recommendations. The 2-week follow-up survey for parents will also re-assess self-efficacy, parental distress, and mental health treatment stigma. The 2-week follow-up survey for youth assesses mood and suicidal thoughts, perceptions of parent support post discharge, and outpatient treatment. It reassesses suicidal risk, depression, connectedness, and alcohol use.
- Phase I (Experimental): Families will complete baseline measures, and receive enhanced usual care from PES clinical staff during their visit as well as a parent toolkit that reinforces evidence-based practices for crisis management such as safety planning and means restriction and encourages parents to increase their support, supervision, and monitoring of their at risk youth. The same follow-up methodology as in Baseline will be utilized.
  Interventions: Behavioral: Parent toolkit; Behavioral: Enhanced Care
- Phase II (Experimental): Families will complete baseline measures and receive Phase I interventions (enhanced care and parent toolkit). Parents will receive caring contacts post discharge, which may occur by phone, text, or email. Caring follow-up messages will provide support, additional education, and problem solving assistance. The same follow-up methodology as in Baseline will be utilized.
  Interventions: Behavioral: Parent toolkit; Behavioral: Enhanced Care; Behavioral: Caring Follow-Up Messages

INTERVENTIONS:
Behavioral: Parent toolkit — The parent tookit is a resource that reinforces evidence-based practices for crisis management such as safety planning and means restriction and encourages parents to increase their support, supervision, and monitoring of their at risk youth.
  Other Names: Toolkit
  Arms: Phase I; Phase II
Behavioral: Enhanced Care — PES clinical staff will receive training on the best practices in brief crisis-focused interventions in emergency settings with parents and youth.
  Arms: Phase I; Phase II
Behavioral: Caring Follow-Up Messages — Parents will receive caring contacts via phone, text, or email to provide support, additional education, and problem solving assistance in the days and weeks post-discharge.
  Other Names: Follow-Up
  Arms: Phase II

SUMMARY:
The Psychiatric Emergency Services (PES) Family Support and Follow-Up Program is a service delivery intervention that utilizes a multi-component approach to enhance usual care provided to youth and families at the University of Michigan Psychiatric Emergency Services in order to promote youth safety and provide support to families following their visit. During the first phase of intervention, families will receive enhanced usual care by clinical staff along with a family toolkit that includes a youth safety plan and written recommendations for safety monitoring and supporting youth during a crisis. During the second phase of intervention, families will receive the interventions provided during the first phase in addition to caring contacts post discharge, which may occur by phone, text, or email. Caring contacts are meant to provide support, additional education, and problem solving assistance.

DETAILED DESCRIPTION:
All participants complete a battery of measures in the waiting room during their PES visit. Youth will complete surveys that collect demographic information, assess current suicidal ideation, perceptions of future suicidal risk, connectedness to others, reasons for living, depression, alcohol use, and self-efficacy. Parents will complete questionnaires that gather demographic information, self-efficacy, baseline means restriction, expectations, hopes, and needs during their visit to PES, assess their child's adaptive functioning and behavioral, social, and emotional adjustment, parent psychiatric history, parental distress, and attitudes about the extent to which seeking mental health treatment is stigmatized. PES clinicians will also administer the Columbia Suicide Severity Rating Scale as part of standard PES practices.

The first phase of intervention (Phase I) involves training clinical staff at PES to implement a new model of service delivery that focuses on the PES visit as an opportunity for crisis intervention for youth and families. The training incorporates best practices in brief crisis-focused interventions in emergency settings. When the provider training is completed, families will receive enhanced usual care by clinical staff along with a toolkit that reinforces evidence-based practices for crisis management such as safety planning, supervision, and monitoring of their at-risk youth. Parents and youth are asked to complete the battery of baseline measures at PES, then an online follow-up survey at 3 days (parents only) and 2 weeks (parents and youth) post discharge. Youth and parents are asked to report on the extent to which they recall their clinician promoting best practice interventions such as safety planning and means restriction during their visit and whether or not they felt their needs were met in PES. Families will also report on barriers accessing outpatient care and need for additional supports. Parents will be asked to report on any means restriction and safety planning activities with their child and whether their child was connected to outpatient services. Youth will be asked to report on the extent to which they feel supported by their families in addition to information about their level of suicide risk.

The second intervention (Phase II) includes the interventions provided during phase I (i.e., enhanced care and toolkit) and caring follow-up contacts for parent participants. Caring contacts post discharge may occur by phone, text, or email. This study will examine the benefit of text messaging contacts in addition to phone contacts in the days and weeks post discharge.

Data from Phase I will be compared to pre-test data obtained at baseline to assess the potential benefits of enhancements to usual care as measured by families' increased abilities to implement safety measures (means restriction, safety plans, risk assessment), support (expressions of caring, modification of expectations), or link their child to outpatient psychiatric treatment. Secondary analyses will explore possible mechanisms of action for family behavior changes (or lack thereof), including levels of parent distress at baseline, parents' stigma regarding receiving psychological services, and markers of the severity of youth psychopathology (i.e., level of suicidality, depression, substance use, functional impairment, and low parental connectedness). Parent ratings of self-efficacy are hypothesized to change with the addition of the interventions during Phase I and Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to U-M Psychiatric Emergency Services
* Experiencing suicide-related concerns

Exclusion Criteria:

* Do not speak English
* Currently experiencing psychosis
* Currently intoxicated
* Cognitively impaired
* Currently experiencing severe aggression or agitation
* Unaccompanied by parent/legal guardian

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 229 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Change in adherence to safety recommendations | Baseline, 3 days, 2 weeks
  Change in the number of families' engaging in safety recommendations including means restriction in the home, safety planning, and risk assessment as measured by yes/no response.
Access to outpatient mental health services | 2 weeks
  The number of youth linked to outpatient mental health services including therapy, psychiatry, or a combination.

SECONDARY OUTCOMES:
Change in parental self-efficacy: Parent Self-Efficacy Form | Baseline, 2 weeks
  Measuring the change in parents' ratings of self-efficacy at baseline and post discharge using the Parent Self-Efficacy Form. This is a 13-item questionnaire developed to assess confidence in promoting safety and talking about suicide with their child. Parents are asked to rate how confident they feel in completing certain actions with their child on a ten-point scale, with 0 being "not confident at all", 5 being "somewhat confident" and 10 being "completely confident." Parents are asked to rate their confidence in performing 13 actions, including asking their child's about his/her mood, identifying suicide warning signs, and completing a safety plan with their child.
Youth connectedness | Baseline, 2 weeks
  Measuring youths' ratings of connectedness at baseline and 2 weeks post discharge using the Parent-Family Connectedness Scale. This is a 13-item self-report measure that assesses the extent to which adolescents feel connected to their parents and family on a 5-point scale. Scale response options include not at all, just a little, somewhat, quite a bit, and very much.
Parental distress | Baseline, 2 weeks
  Measuring parental distress using the Pediatric Inventory for Parents. This questionnaire was developed to measure the stress of caring for a child with an illness and was initially validated among pediatric oncology populations. The measure has been adapted to measure the stress of parenting a child experiencing high suicidality. The instrument asks the respondent to indicate the frequency and difficulty of 34 events over the past 7 days using a 5-point scale. Response options for frequency include never, rarely, sometimes, often, and very often. Response options for difficulty include not at all, a little, somewhat, very much, and extremely. The instrument is scored separately for each of the 3 domains: Communication (range: 8-40), Emotional Distress (range: 15-75), and Role Function (range: 10-50). Higher scores indicate higher levels of distress.
Youth suicidality | Baseline, 2 weeks
  Measuring youth suicidality at baseline and 2 weeks post discharge using the Suicidal Ideation Questionnaire-Junior. The SIQ-JR is a 15-item questionnaire that assesses the frequency of suicidal ideation. It is scored on a 0-6 scale, and a cutoff score of 31 is considered optimal to identify youth at higher risk.
Parent stigma for receiving psychological help | Baseline, 2 weeks
  Measuring parents' attitudes about the extent to which seeking mental health treatment is stigmatized at baseline and 2 weeks post discharge using the Stigma Scale for Receiving Psychological Help. This survey includes 5 items, each rated on a 4-point Likert scale, ranging from 0 (Strongly Disagree) to 3 (Strongly Agree). It has been slightly modified for this study by changing the exclusive focus on "psychological treatment." The word "psychologist" has been replaced by mental health professional.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ewell Foster, Ph.D., Principal Investigator — University of Michigan; Patricia Smith, MA, Principal Investigator — Michigan Department of Health and Human Services
Locations (1):
- University of Michigan Psychiatric Emergency Services, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No